CLINICAL TRIAL: NCT02998281
Title: Effects of Inspiratory Muscle Training on Respiratory Functions, Trunk Control, Activities of Daily Living, Functional Exercise Capacity and Quality of Life in Children With Cerebral Palsy
Brief Title: Effects of Inspiratory Muscle Training in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Muserrefe Nur Keles, MSc Pt, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1234
Record Dates: First submitted 2016-12-10; First posted 2016-12-20 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Cerebral Palsy; Respiration; Decreased
Keywords: cerebral palsy; inspiratory muscle training
MeSH Terms: conditions — Cerebral Palsy; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Active Comparator): The treatment group received Inspiratory muscle training (IMT) at 40% of maximal mouth pressure (PImax) by using Threshold IMT and training loads were adjusted to maintain 40% of the PImax weekly. The PImax was measured at supervised sessions each week, and 40% of the measured value was determined as the new training work load.
  Interventions: Device: Threshold (IMT)
- Control Group (Sham Comparator): The control group received sham Inspiratory muscle training (IMT) at a fixed work load, 5% of PImax by using Threshold IMT.
  Interventions: Device: Threshold (IMT)

INTERVENTIONS:
Device: Threshold (IMT) — Training is going to perform by using a pressure threshold- loading device (Threshold, IMT, USA) used to inhale against a same-pressure load every inhalation for strengthening primarily the diaphragm and rib cage muscles. The device pressure is adjusted according to PImax, and reliability/reproducibility has been demonstrated.

SUMMARY:
Even if cerebral palsy not directly effect respiratory system, impairment of nervous and muscle systems, because of the brain damage, may cause respiratory functions impairment. In literature, it has been showed that children with cerebral palsy have decreased respiratory muscle strength and associated with trunk control, quality of life and respiratory functions. But, there is no study in literature that aims to increase respiratory muscle strength in these children. Hence, the aim of this study is to investigate effects of inspiratory muscle training on respiratory functions, trunk control, activities of daily living, functional exercise capacity and quality of life in children with cerebral palsy.

DETAILED DESCRIPTION:
A convenience of children with hemiparetic and diplegia CP, 7-14 years, is going to recruited from Gazi University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation. Patients will randomly allocate to either a treatment group or control group. The treatment group will receive inspiratory muscle training at 30-40% of maximal mouth pressure, the control group will receive sham inspiratory muscle training at a fixed work load, 5% of maximal mouth pressure. Groups are going to train for a total of 30 min/d, 7 days/week, for 6 weeks. Before and after treatment, every each of patients pulmonary function test will be evaluated with using spirometry, respiratory muscle strength using with electronic mouth pressure device, trunk control with using trunk control measurement scale, activities of daily living using with Pediatric Evaluation of Disability Inventory (PEDI), functional exercise capacity usin with six minute walk test (6MWT) and quality of life using with Cerebral Palsy Quality of Life Questionnaire (CPQOL).

ELIGIBILITY:
Inclusion Criteria:

* Aged 7-14 years
* Diagnosed to spastic cerebral palsy
* Gross Motor Function Classification System levels I or II.
* Have no earlier interventions in the form of orthopaedic surgery or injection with botulinum toxin type A in the 6 month prior to baseline assessments
* Child are able to demonstrate sufficient co-operation and cognitive understanding participating

Exclusion Criteria:

* Active medical condition impairment (pneumonia etc.)
* Do not accommodate the study
* Do not want to attempt the study

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2016-12; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test | 6 weeks
  this is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair and sit down. During the test, the child is expected to wear their regular footwear and use any mobility aids that they would normally require.

SECONDARY OUTCOMES:
Activities of daily living using with Pediatric Evaluation of Disability Inventory | 6 weeks
  PEDI scale
Pulmonary Function Test | 6 weeks
  spirometry
Respiratory muscle strength | 6 weeks
  Mouth pressure device
Functional exercise capacity | 6 weeks
  six minute walk test
Change in trunk control over time assessed with Trunk Control Measurement Scale | 6 weeks
  Assessing change in trunk control

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Elbasan, Phd, Study Chair — Gazi University
Locations (1):
- Gazi University, Faculty of Health and Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We have no decided yet